CLINICAL TRIAL: NCT07113015
Title: Comparative Efficacy and Safety of Propranolol Versus Amantadine in Controlling Tremors in Parkinson's Disease: A Randomized Controlled Trial
Brief Title: A Study Comparing Propranolol and Amantadine for Reducing Tremors in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Multan Medical And Dental College (Other)
Responsible Party: Principal Investigator, Nabeel Ahmed, Principal Investigator, Multan Medical And Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MultanMDC1
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease (PD); Tremor
Keywords: Amantadine; Parkinson's Disease; Propranolol; Motor Symptoms; Tremors
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — Propranolol; Amantadine; GluN2C-2D antagonist UBP145

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Propranolol (Active Comparator): Received 40 mg of propranolol administered orally twice daily, with dose titration permitted based on clinical response and tolerability, not exceeding 80 mg/day. PD medications remained unchanged during the trial.
  Interventions: Drug: propranolol
- Group Amantadine (Active Comparator): Received 100 mg of amantadine administered orally twice daily, with dose titration permitted based on clinical response and tolerability, not exceeding 200 mg/day. PD medications remained unchanged during the trial.
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: propranolol — 40 mg orally twice daily, titrated up to a maximum of 80 mg/day.
  Other Names: Inderal; Non-selective beta-blocker
  Arms: Group Propranolol
Drug: Amantadine — 100 mg orally twice daily, titrated up to a maximum of 200 mg/day.
  Other Names: Symmetrel; NMDA receptor antagonist
  Arms: Group Amantadine

SUMMARY:
Parkinson's disease is a common brain disorder in older adults that causes tremors (shaking), stiffness, and problems with movement. Among these symptoms, tremors-especially those that occur at rest-can be distressing and interfere with daily life. This study aims to compare two commonly used medications, propranolol and amantadine, to determine which one is more effective and safer in reducing tremors in people with Parkinson's disease.

This clinical trial was conducted with 220 adults aged 50 to 80 years who had a confirmed diagnosis of Parkinson's disease and noticeable resting tremors. Participants were randomly assigned to receive either propranolol or amantadine for 12 weeks, while continuing their usual Parkinson's medications. Tremor severity was measured using a standard scoring tool known as the Unified Parkinson's Disease Rating Scale (UPDRS). Quality of life and side effects were also closely monitored.

The hypothesis is that propranolol would be more effective in reducing tremor severity than amantadine, though it might be associated with more side effects. Both medications were given in tablet form, twice daily, and doses were adjusted based on patient response and tolerance.

At the end of the study, both groups showed improvement, but propranolol was more effective at reducing tremors. However, it caused more side effects such as tiredness and dizziness. Quality of life improved in both groups with no major difference between them. This study may help doctors decide which medication is more suitable for treating tremors in Parkinson's disease, based on the patient's health status and side effect tolerance.

ELIGIBILITY:
Inclusion Criteria:

* UK Parkinson's Disease Society Brain Bank criteria [7] - Parkinson's Disease.
* Aged between 50 and 80 years.
* Significant (resting tremor score, defined as η ≥2 on the UPDRS Part III).
* At least 4 weeks prior to the study, a stable regimen of PD medication.

Exclusion Criteria:

* Severe bradycardia, history of asthma, or heart block (used instead of the propranolol group).
* History of seizures or significant renal impairment (Amantadine group).
* Cigarette smoking, pregnant or breastfeeding women.
* Patients with MMSE < 24.
* Participation in another clinical trial at the same time.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Change in tremor severity | From baseline to 12 weeks after intervention initiation
  This measure assessed the severity of resting tremor using Part III (Motor Examination) of the Unified Parkinson's Disease Rating Scale (UPDRS). Each tremor item was scored from 0 to 4, with higher scores reflecting greater severity. The change in tremor scores from baseline to week 12 was used to evaluate and compare the efficacy of propranolol and amantadine in reducing tremor severity among participants with Parkinson's disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Multan Medical and Dental College, Multan, Punjab Province, Pakistan